CLINICAL TRIAL: NCT00003469
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Children With Rhabdoid Tumor of the Central Nervous System
Brief Title: Antineoplaston Therapy in Treating Children With Rhabdoid Tumor of the Central Nervous System
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066505; BC-BT-14 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Rhabdoid Neoplasm of CNS
Keywords: childhood rhabdoid tumor
MeSH Terms: conditions — Rhabdoid Tumor | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Children with a Rhabdoid tumor will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for childhood Rhabdoid tumors provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of childhood Rhabdoid tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children (> 6 months of age) with Rhabdoid tumors.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which children with Rhabdoid tumors receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in children with a Rhabdoid tumor, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in children with a Rhabdoid tumor.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Rhabdoid tumor of the central nervous system that is unlikely to respond to existing therapy and for which no curative therapy exists
* Measurable tumor by MRI scan performed within two weeks prior to study entry
* Tumor must be at least 5 mm

PATIENT CHARACTERISTICS:

Age:

* 6 months to 17 years

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No severe heart disease
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concomitant disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on a stable dose for at least 1 week before study entry)

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston treatment

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 1996-02; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four patients were recruited between February 1996 and May 2003. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: Years] | 3.7 [2.0 to 6.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 4
Participants
  Partial Response | 1
  Stable Disease | 1
  Progressive Disease | 2

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months overall survival
Time Frame: 6 months, 12 months, 24 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 4
Percentage of participants
  6 months overall survival | 75.0
  12 months overall survival | 50.0
  24 months overall survival | 0.0

ADVERSE EVENTS:
Time Frame: 7 years, 2 months
Description: Four patients were recruited between February 1996 and October 2010. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=4)
Central Venous Catheter Infection (General disorders) | 1 — The Central Venous Catheter Infection was not related to Antineoplaston therapy
Vomiting (Gastrointestinal disorders) | 1 — The Vomiting was not related to Antineoplaston therapy
Hypernatremia (Investigations) | 1 — The Hypernatremia was not related to Antineoplaston Therapy.
Hypokalemia (Investigations) | 1 — The Hypokalemia was not related to Antineoplaston therapy.
Pain: Head/headache (Nervous system disorders) | 1 — The Pain: Head/headache was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=4)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Hypotension (Cardiac disorders) | 1
Central venous catheter infection (Infections and infestations) | 1
Non-functional central venous catheter (General disorders) | 2
Fatigue (asthenia, lethargy, malaise (General disorders) | 2
Fever (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Infection (documented clinically): Sinus (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Hypernatremia (Investigations) | 3
Hyperuricemia (Investigations) | 1
Hypoglycemia (Investigations) | 1
Hypokalemia (Investigations) | 4
Hypomagnesemia (Investigations) | 1
Uric acid, serum-high (hyperuricemia) (Investigations) | 1
Neuropathy: motor (Nervous system disorders) | 1
Speech impairment (Nervous system disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Pain: Head/headache (Nervous system disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Flu-like syndrome (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No